CLINICAL TRIAL: NCT03638765
Title: A Phase Ib Clinical Trial Evaluating DCVax-Direct, Autologous Activated Dendritic Cells for Intratumoral Injection, in Patients With Unresectable Brain Metastases From Breast- or Non-Small Cell Lung Cancer
Brief Title: Dendritic Cell Therapy for Brain Metastases From Breast- or Lung Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Northwest Biotherapeutics (Industry)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 050811
Record Dates: First submitted 2018-08-15; First posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Brain Metastases; Lung Cancer Metastatic; Breast Cancer Metastatic
Keywords: immunotherapy; dendritic cells; brain metastases
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental Treatment (Experimental): Intratumoral injection of activated, autologous dendritic cells (DCVax-Direct) in brain metastases from lung cancer or breast cancer
  Interventions: Biological: DCVax-Direct

INTERVENTIONS:
Biological: DCVax-Direct — activated, autologous dendritic cells

SUMMARY:
The study will use an Ommaya reservoir that drains into brain metastases to deliver activated, autolous dendritic cells to the tumor lesion, for patients who are 18 - 75 years old who have brain metastases from either lung cancer or breast cancer. The primary objective of the study is to evaluate the safety and feasibility of administering DCVax-Direct to patients with metastatic tumors in the brain. The secondary objectives are to determine tumor response, the rate of intracranial recurrence (IR), the rate of neurologic deaths, decline in neuro-cognitive functioning and overall survival. Approximately 10 patients with injectable metastatic brain tumors will be enrolled initially in a dose escalation scheme, with the expectation to enroll a total of 24 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent
2. Age between 18 and 75 years (inclusive) at screening.
3. Willingness to provide Social Security Number to facilitate survival follow up.
4. Pathologically confirmed metastatic breast or non-small cell lung cancer
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1 or 2
6. Adequate bone marrow function, as indicated by the following:
7. Adequate renal function
8. Adequate liver function
9. Life expectancy > 12 weeks
10. Negative serum pregnancy test done ≤7 days prior to registration, for women of childbearing potential only.
11. Determined prior to enrollment: sufficient number of doses of DCVax-Direct manufactured to complete 7 injections. A second leukapheresis is allowed to meet this requirement if necessary.
12. Unequivocal evidence of newly diagnosed untreated brain metastases and/or progressive brain metastases after previous whole brain radiation therapy (WBRT), currently amenable to stereotactic radiosurgery
13. At least one CNS metastasis accessible for reservoir placement
14. At least one measurable CNS metastasis (lesion ≥ 10 mm per RANO-BM criteria)

Exclusion Criteria:

1. Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm OR Participated in a study of an investigational agent, received study therapy or used an investigational device ≤4 weeks prior to registration
2. Immunocompromised patients and patients with known immunodeficiency
3. Patients receiving systemic steroid therapy >10 mg prednisone or equivalent or any other immunosuppressive therapy ≤7 days prior to registration. NOTE: Inhaled steroids and low-dose corticosteroids are allowed.
4. History of active tuberculosis (TB), human immunodeficiency virus (HIV), active hepatitis B (e.g., HBsAg reactive) and/or active hepatitis C infection (e.g. HCV RNA qualitative is detected).
5. Active autoimmune disease requiring systemic treatment in the past 2 years (i.e. use of disease modifying agents, corticosteroids or immunosuppressive drugs). NOTE: Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
6. Known history of, or any evidence of active, non-infectious pneumonitis.
7. Active infection requiring systemic therapy.
8. Other active malignancy ≤3 years prior to registration. EXCEPTIONS: Adequately treated non-melanotic skin cancer (adequate wound healing is required prior to study entry) or carcinoma-in-situ of the cervix. NOTE: If there is a history of prior solid tumor malignancy, it must have been treated curatively with no evidence of recurrence ≤3 years prior to registration.
9. Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g., infection/inflammation, intestinal obstruction, unable to swallow medication, social/ psychological issues, etc.
10. Medical, psychiatric, cognitive or other conditions that may compromise the patient's ability to understand the patient information, give informed consent, comply with the study protocol or complete the study.
11. Stage IV lung cancer patients with actionable EGFR, ALK or ROS-1 alteration will be excluded from the study.
12. Serious medical conditions
13. Any systemic myelotoxic chemotherapy within 8 weeks prior to screening
14. Evidence of recent hemorrhage on MR at pre-screening
15. Positive HIV-1, HIV-2, or HTLV-I/II tests.
16. History of multiple sclerosis
17. Requirement for ongoing immunosuppressants
18. Ongoing medical need for continuous anti-coagulation or anti-platelet medication,
19. Known genetic cancer-susceptibility syndromes such as Li-Fraumeni syndrome
20. Ongoing fever for longer than 48 hours of ≥ 101.5oF/38.6oC at screening
21. Females of child-bearing potential who are pregnant or lactating or who are not using adequate contraception.
22. Allergy or anaphylaxis to any of the reagents used in this study
23. Inability or unwillingness to return for required visits and follow-up exams

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Safety is assessed graded according to NCI CTC. The overall incidence of adverse events is calculated. | Through study completion, an average of 6 months
  Toxicity is monitored and graded according to NCI CTC. The overall incidence of adverse events is calculated

SECONDARY OUTCOMES:
tumor response | Every 8 weeks through study completion, an average of 6 months
  Tumor response is assessed through radiographic means and must at a minimum include MRI scans with and without contrast. The newly proposed iRANO criteria are used to characterize responses
intracranial recurrence rate | Every 8 weeks through study completion, an average of 6 months
  Tumor recurrence in the brain is assessed through radiographic means and must at a minimum include MRI scans with and without contrast. The newly proposed iRANO criteria are used to characterize recurrences
overall survival | Through study completion, an average of 6 months
  Time to death for each subject, measured from time of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Quinones Hinojosa, MB, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No